CLINICAL TRIAL: NCT03788902
Title: Oxytocin and Social Cognition in Children With Attention Deficit Hyperactivity Disorder: Impact of Methylphenidate
Brief Title: OT and Social Cognition in Children With ADHD: Impact of MPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Principal Investigator, Yuval Bloch, Head of child and adolescent outpatient clinic, Shalvata Mental Health Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 0017-13-SHA
Record Dates: First submitted 2018-12-19; First posted 2018-12-28 (Actual); Last update posted 2018-12-28 (Actual); Status verified 2018-12

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ADHD group (Experimental): This group was examined twice - once after taking Ritalin and once after taking placebo
  Interventions: Drug: Ritalin
- Healthy control (No Intervention): Children with the same demographics as children with ADHD but without ADHD or a first degree relative with ADHD

INTERVENTIONS:
Drug: Ritalin — Single dose of Ritalin IR 0.3-0.5 mg/kg OR placebo
  Arms: ADHD group

SUMMARY:
Background: The current study aimed to explore the possible effect of stimulants on oxytocin (OT), a neuropeptide found to regulate social behavior, as a mediator of the pro-social effect of methylphenidate (MPH) in children with attention deficit hyperactivity disorder (ADHD) compared to healthy controls (HCs). Methods: In a double-blind manner the investigators compared the performance of 50 children with ADHD and 40 HCs in "theory of mind" (ToM) tasks and examined the effect of a single dose of MPH/placebo on ToM and salivary OT levels in children with ADHD at baseline and following an interpersonal interaction.

DETAILED DESCRIPTION:
Attention deficit hyperactivity disorder (ADHD), a neurodevelopmental disorder affecting approximately 7% of children and adolescents, is associated with considerable impairments in social functioning. Children with ADHD, in comparison to healthy children, suffer from more social rejection and problems in reciprocal relationships. Deficits in interpersonal functioning in children with ADHD have been attributed in previous studies to, among other things, impairments in theory of mind (ToM) - the ability to attribute mental states, beliefs, and intentions to self and to others. For example, some studies have shown deficits in the ability to recognize facial expressions among children with ADHD. Other studies have found impairments in first- and second-order ToM tests. There is also evidence showing that empathic functions in children with ADHD are impaired. However, small sample sizes, as well as high percentages of comorbid disruptive disorders, served as limitations in these studies.

One's ToM ability depends on, among other things, the integrity of dopaminergic and serotonergic systems, as well as on their interaction with other neurotransmitters and neurohormones (e.g., acetylcholine, oxytocin).

Oxytocin (OT) is a neuropeptide found to accelerate the formation of social relationships, the expression of behaviors of closeness, and the recognition of affect in the facial expressions of others. Oxytocin has been hypothesized to raise the salience of social cues by modulating attention-orienting responses to external contextual social cues. Its secretion increases in response to interpersonal interactions. Studies found connections between blood and saliva OT levels, OT receptor gene polymorphism, and the strength of social relationships and behaviors in healthy individuals, as well as in patients suffering from mental disorders. Oxytocin reciprocally interacts with dopaminergic neurons in the mesolimbic tract. Anatomical and immonucytochemical studies have found that neuronal fibers and receptor binding-sites of OT and dopamine are located in the same areas in the central nervous system (CNS), sometimes in very close proximity to one another. Oxytocin-secreting cells in the hypothalamus carry dopamine receptors. Indeed, patients with mental disorders related to dysregulation of dopamine (e.g., autistic spectrum disorders, schizophrenia, depression) show changes in their CNS and peripheral OT levels. Given the fact that injury of dopaminergic transporters and receptors is a central component in the etiology of ADHD, it is also possible that OT plays a role as a mediator of social deficits, and mainly in ToM impairment in children with ADHD.

To date, only a few studies have shown decreased OT levels in children with ADHD when compared to healthy controls. These studies found a negative correlation between serum OT levels and ADHD rating scale total scores, and aggression scores, and a positive correlation between the serum OT level and empathy scores in patients with ADHD. However, in both studies, only baseline OT levels were assessed; therefore, changes in OT levels following an interpersonal interaction were not measured. This is an important point, as social abilities are dynamic and interaction-related; the reactivity of the OT system to interpersonal interaction is thus probably highly relevant to the understanding of social difficulties in ADHD patients.

Stimulants reduce negative social interactions and improve social and behavioral functioning in children with ADHD, and also improve empathy scores. In a previous study, the investigators showed that a single dose of methylphenidate (MPH) improved the performance of children with ADHD on ToM tests. To date, no study examined a possible effect of stimulants on OT levels in children with ADHD. This is a pivotal issue in the understanding of the neurobiological underpinnings of improvement in social cognition measures among children with ADHD who are treated with stimulants, given that OT might have a role in mediating this improvement.

In the current study the investigators hypothesized that dysfunction in the OT system may account for the social difficulties of children suffering from ADHD and that the dynamics in the OT system may explain the pro-social effect of stimulants on these children. Thus, the objectives of the current study were 1) to compare ToM measures and salivary OT levels between children with ADHD and healthy controls (HCs), and 2) to examine the effect of a single dose of MPH on ToM and salivary OT levels in children with ADHD following an interpersonal interaction.

Methods Subjects Fifty children aged 6-12 diagnosed with ADHD and 40 HCs were recruited. Patients were recruited from the ADHD clinic and the outpatient clinic of the Shalvata Mental Health Center, School of Medicine, Tel-Aviv University. The HCs subjects were recruited from the community via the internet and social media.

ADHD was diagnosed by child and adolescent psychiatrists using the Diagnostic and Statistical Manual of Mental Disorders, fourth or fifth edition (DSM-IV-TR and DSM-5). The investigators excluded children with a past or current affective disorder, psychosis, substance abuse, conduct disorder or any medical or neurological condition or medication-taking that might affect the child's participation in the study. The investigators also excluded children who had a first-degree relative with a major psychiatric diagnosis.

Inclusion criteria for the control group were the same as those of the ADHD group but with no diagnosis of ADHD or a first-degree relative with ADHD.

Participants were reimbursed for their expanses in participation and received a small present as appreciation. The IRB approved the study. Both parents of all participants signed a consent form and the children gave their consent verbally.

Procedure Apart from the initial clinical assessment at the clinic, all assessments were performed in the children's homes. Children with ADHD participated in two sessions: one session an hour after taking a short-acting MPH (in an adjusted dosage of 0.3-0.5mg/kg) and one session an hour after taking a placebo (PLC). Children routinely prescribed with MPH treatment were asked not to take the medicine 48 hours before the examination, since the clinical effect of the long-acting MPH is no longer than 12 hours. The study was randomized-controlled, such that children were assigned to the sessions randomly in a double-blind manner. Each session lasted about 60-90 minutes. In order to lessen a possible learning effect of the computerized tasks (to be elaborated upon forthwith), the sessions were performed at least two weeks apart. Control subjects participated in only one session and did not take any medication.

Parents completed questionnaires regarding demographics and general information about the child's academic and social functioning. In addition, parents completed the Swanson, Nolan and Pelham Questionnaire-IV (SNAP-IV). This instrument contains subscales for inattention, hyperactive/impulsive behavior, and oppositional behavior.

Parents also filled out the Strengths and Difficulties Questionnaire (SDQ), a screening inventory composed of five distinct dimensions: conduct problems, emotional symptoms, hyperactivity, peer problems, and pro-social behavior. Intelligence was measured using the similarities subtest from the Wechsler Intelligence Scale for Children version IV (WISC-IV). Self-reported anxiety was measured using the State-Trait Anxiety Inventory (STAI), a 40-item questionnaire scored by a Likert scale. State anxiety represents a transient emotional status that results from situational stress; trait anxiety represents a predisposition to react with anxiety in stressful situations.

The investigators measured ToM performance using the ToM test, which test consists of vignettes, stories, and drawings about which the child has to answer a number of questions. Results are given on three subscales: ToM1 - precursors of ToM (i.e., recognition of emotions); ToM2 - first manifestations of a real ToM (first-order belief, understanding of false belief); and ToM3 - more advanced aspects of ToM (second-order belief, understanding of humor). The second ToM task was the Faux Pas Recognition task (FPR), designed by Baron-Cohen et al.. This task is designated to evaluate the ability of participants to recognize social "faux pas" - social situations in which a speaker says something without understanding that there might be a difference between his/her state of knowledge and that of the listener ("cognitive" ToM), and should recognize the potential emotional impact of a statement on the listener ("affective" ToM). At each session, participants were given 10 short stories, five of which contained faux pas situations to be identified. After hearing every story, participants were asked ToM questions. The score consisted of the total number of all correct identifications of a faux pas situation. The Hebrew version of the FPR was employed after validation by a group of normative subjects.

Executive functions and attention were tested via the cognition module in the NIH Toolbox for the Assessment of Neurological and Behavioral Function (NIH-TB). The investigators used the Dimensional Change Card Sort Test (DCCS) and the Flanker Inhibitory Control and Attention Test, which measure cognitive flexibility and inhibitory control, respectively.

Salivary OT levels were measured at three time points: at the beginning of each session ("T1"), 40 minutes after the administration of MPH/PLC ("T2"; only for the ADHD group), and 15 minutes after a "positive social interaction" in which the child and the parent were asked to plan a "fun day" that would include both of them, and to talk about it for five minutes ("T3"). Participants were asked to avoid drinking and eating an hour before the test and to avoid caffeine three hours before the test.

Saliva samples were collected by passive drool. In order to precipitate the mucus, samples underwent three freeze-thaw cycles: freeze at -70°C and thaw at 4°C. After the forth cycle the tubes were centrifuged twice at 1500 x g (4000 rpm) for 30 minutes. Supernatants were collected and stored at -20°C until assayed. Determination of OT from saliva samples was performed using a commercial OT ELISA kit (ENZO, NY, USA). Measurements were performed in duplicate according to the manufacturer's instructions. The concentrations of samples were calculated using MatLab-7 according to relevant standard curves. The intra-assay and inter-assay coefficients of samples were 14.7 and 22.7 percent, respectively. The intra-assay and inter-assay coefficients of controls were 4.9 and 13.2 percent, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Ages 6-12 years
* Diagnosis of ADHD

Exclusion Criteria:

* Past or current affective disorder, psychosis, substance abuse, conduct disorder
* Any medical or neurological condition or medication-taking that might affect the child's participation in the study
* First-degree relative with a major psychiatric diagnosis

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
changes in scores of ToM test | 20 minutes
  ToM test - consists of vignettes, stories, and drawings about which the child has to answer a number of questions.
changes in scores of Faux-Pas Recognition test | 15 minutes
  number of faux-pas recognized in specific vignettes by participants
changes in Oxytocin salivary level | 2 hours
  Oxytocin salivary levels as measured three/two times during the examination (ADHD group and healthy control accordingly).

CONTACTS AND LOCATIONS:
Overall Officials: Hagai Maoz, MD, Principal Investigator — Shalvata Mental Health Center

IPD SHARING:
Plan to Share IPD: No